CLINICAL TRIAL: NCT02833597
Title: Claudication Evaluation During Rowing ExerciseS. Rehabilitation Arteritis of Lower Limbs by Rowing
Brief Title: Claudication Evaluation During Rowing ExerciseS
Acronym: CERES
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2015-A00189-40
Record Dates: First submitted 2016-06-14; First posted 2016-07-14 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Peripheral Artery Disease
Keywords: peripheral artery disease; transcutaneous oxygen pressure; claudication; rowing ergometer
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Check the feasibility of the collection of reliable measures of tcpO2 the lower limbs in arteriopathy when performing rowing on effort.

DETAILED DESCRIPTION:
Obtaining curve values of tcpO2 interpretable when recording the effort by rowing on rowing.

Show the occurrence of ischemia in the lower limbs during recording effort by rowing on rowing

ELIGIBILITY:
Inclusion Criteria:

* referred for an oximetry exercise test
* Patient able to walk on a treadmill
* Patient covered by the French health insurance
* Patient able to understand the protocol
* Patient agrees to be involve in the protocol and sign the consent form

Exclusion Criteria:

* any heart issues during the last 3 months
* pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with buttock pain and referred for an oximetry exercise test
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2016-07; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Changes in transcutaneous oxygen pressure (tcpo2) value in the calf for different rowing intensities | up to 1 day
  during exercise on rowing ergoùmeter, we collect reliable measurements of TcPO2 on chest and limb and calculate the DROP index (Limb changes minus chest changes)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre ABRAHAM, MD; Ph.D, Principal Investigator — University hospital, Angers, FRANCE
Locations (1):
- University Hospital, Angers, France

IPD SHARING:
Plan to Share IPD: No